CLINICAL TRIAL: NCT04016389
Title: FIGO 2018 Stage IB2 (> 2 to ≤4cm) Cervical Cancer Treated With Neoadjuvant Chemotherapy Followed by Fertility Sparing Surgery (CoNteSSa) / Neo-Adjuvant Chemotherapy and Conservative Surgery in Cervical Cancer to Preserve Fertility
Brief Title: FIGO 2018 Stage IB2 Cervical Cancer Treated With Neoadjuvant Chemotherapy Followed by Fertility Sparing Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hotel Dieu Hospital (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CoNteSSa; CoNteSSa - NeoCon (Other: Princess Margaret Cancer Centre); NCT04483557 (obsolete NCT alias)
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Carboplatin; Paclitaxel; Trachelectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neo-Adjuvant Chemotherapy, Surgery, and Adjuvant Chemotherapy (Experimental): Participants will receive neo-adjuvant treatment cisplatin or carboplatin with paclitaxel, intravenously, either once every cycle or once a week, for three (21-day) cycles.
  After neo-adjuvant treatment, depending on their status, participants may have the trachelectomy done.
  Adjuvant treatment may include standard chemotherapy and radiotherapy, or a hysterectomy may need to be done.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Trachelectomy

INTERVENTIONS:
Drug: Cisplatin — Cisplatin is an antineoplastic agent that is commonly used for the treatment of cervical cancer.
Drug: Carboplatin — Carboplatin is an antineoplastic agent that is commonly used for the treatment of cervical cancer.
Drug: Paclitaxel — Paclitaxel is an antineoplastic agent that is commonly used in combination with cisplatin or carboplatin for the treatment of cervical cancer.
Procedure: Trachelectomy — Surgery to remove the cervix but keep the uterus intact.

SUMMARY:
This study will include patients with invasive cervical cancer that wish to keep their fertility as much as possible in the future after treatment.

Patients who receive surgery alone may experience long-term side effects including infertility. The purpose of this research study is to determine whether giving neo-adjuvant chemotherapy prior to surgery can maintain fertility in patients with invasive cervical cancer.

The neo-adjuvant chemotherapy will consist of a platinum-based chemotherapy drug cisplatin or carboplatin, with a chemotherapy drug called paclitaxel. These are common chemotherapy drugs used in the treatment of women with cervical cancers.

DETAILED DESCRIPTION:
All participants will first receive neo-adjuvant platinum-based chemotherapy. Once the neo-adjuvant chemotherapy has been completed, participants will be assessed by imaging scans to see whether they have a response to the treatment.

If participants are responding to treatment, they will then have a trachelectomy. After surgery, participants will be assessed and the study doctor will determine whether adjuvant treatment is needed. Adjuvant treatment may include chemotherapy and radiotherapy, or have a hysterectomy done.

If participants do not respond to or their disease worsens after neo-adjuvant treatment, participants will receive adjuvant treatment with chemotherapy and radiotherapy or have a hysterectomy done.

ELIGIBILITY:
Inclusion Criteria:

Part 1 - Eligibility Criteria for Neoadjuvant Chemotherapy

* Patients must have histologically confirmed invasive cervical cancer with adenocarcinoma, adenosquamous or squamous histology and FIGO 2018 IB2 measuring >2 cm - ≤4 cm by radiological imaging (MRI).
* Patients must be premenopausal and wish to preserve fertility.
* At time of registration, patient may not have had any prior therapy to treat their cancer lesion.
* Eastern Cooperative Group (ECOG) performance status ≤ 2.
* Within 7 days of the proposed start of treatment, patients must have normal organ and marrow function.
* No evidence of active uncontrolled infection (patients on antibiotics are eligible).
* Patient must have disease that is measurable per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Ability to understand and willing to sign a written informed consent document.
* Patients must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least one year after the fertility-sparing surgery (FSS) procedure. A serum pregnancy test within 72 hours prior to study registration is required.

Part 2 - Eligibility Criteria for Fertility Sparing Surgery (FSS)

* Completed 3 cycles of neo-adjuvant chemotherapy and achieved a complete response (CR) or partial response (PR) with reduction of the lesion to <2 cm on physical examination and MRI.

Exclusion Criteria:

Part 1 - Exclusion Criteria for Neoadjuvant Chemotherapy

* Patients who have had chemotherapy or radiotherapy or surgery for their cancer.
* Patients who are receiving any other investigational agents.
* Patients with other cancers requiring ongoing treatment.
* Patients with known / evidence of brain metastases are excluded from participation in this clinical trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel, carboplatin, or cisplatin or other agents used in study.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues.

Part 2 - Exclusion Criteria for Fertility Sparing Surgery

* Patient unable to complete 3 cycles of neoadjuvant chemotherapy
* Suboptimal response to neoadjuvant chemotherapy according to investigator
* Residual lesion > 2cm or disease progression while on chemotherapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of functional uterus defined as successful fertility sparing surgery (FSS) with no adjuvant therapy | 2 years

SECONDARY OUTCOMES:
Number of side effects | 2 years
  By Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Rate of completion of neo-adjuvant chemotherapy | 2 years
Response rate following neo-adjuvant chemotherapy | 2 years
  By Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Rate of fertility sparing surgery | 2 years
Surgical complication rate following fertility sparing surgery | 2 years
  By Clavien-Dindo classification of surgical morbidity
Rate of recurrence-free survival | 2 years
Rate of recurrence-free survival | 3 years
Overall survival for patients who undergo neo-adjuvant chemotherapy followed by fertility sparing surgery | 2 years
Overall survival for patients who undergo neo-adjuvant chemotherapy followed by fertility sparing surgery | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (4):
- MD Anderson Cancer Centre, Houston, Texas, United States
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - L'Hôtel-Dieu de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No